CLINICAL TRIAL: NCT03889990
Title: Acute Effects of a Heat-not-burn Tobacco Product on Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Athanasia Pataka, Assistant Professor of Respiratory Medicine, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8/22.2.2017, 369
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Heated Tobacco; Respiratory Function; Tobacco Toxicity
Keywords: pulmonary function; IQOS; heated tobacco
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy smokers (Other): Healthy smokers males, aged >18years, with >10 pack/years,receiving no medications
  Intervention: the use of an IQOS
  Interventions: Device: IQOS

INTERVENTIONS:
Device: IQOS — "Smoke" IQOS

SUMMARY:
Background: IQOS ("I-Quit-Ordinary-Smoking,") is a type of the growing class of "heat-not-burn" (HNB) tobacco products. The effect of the acute exposure to IQOS smoke on the pulmonary function of healthy smokers has not been studied extensively.

Objectives: Evaluation of the acute effects of IQOS on pulmonary function.

Methods: Healthy non symptomatic smokers, underwent exhaled CO measurement, spirometry including flows, volumes and diffusion capacity, and measurement of their respiratory resistances at 5, 10 and 20 Hz (R5Hz, R10Hz and R20Hz) with the use of an impulse oscillometry system (IOS) before and 15 min after the use of an IQOS.

DETAILED DESCRIPTION:
All participants underwent pulmonary function tests (PFT) (MasterScreen PFT, Jaeger, Wurzburg, Germany) and total respiratory resistances measurement with an impulse oscillometry system (IOS)( (Viasys Jaeger MasterScreen IOS system).From the basic pulmonary measurements (flows and dynamic lung volumes), Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), Tiffenau index (FEV1/FVC, FEV1%), Peak Expiratory Flow (PEF), Maximal Expiratory Flow (MEF) at 25%, 50%, and 75% of vital capacity, Functional Residual Capacity (FRC), Total Lung Capacity (TLC), Residual Volume (RV), Diffusion Capacity (DLCO) were measured. Each manoeuvre was repeated for at least three technically acceptable forced expiratory flow curves in order to attain the best results. Respiratory impedance at 5 Hz (Z5Hz) and respiratory resistance at 5, 10, and 20 Hz (R5Hz, R10Hz, and R20Hz, respectively), reactance at 5, 10, and 20 Hz and resonant frequency were assessed with IOS.

After smoking heated tobacco (IQOS): 5 minutes after smoking IQOS , they repeated again PFTs and IOS measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy smokers,
2. >10 pack/years
3. receiving no medications
4. no co morbidity

Exclusion Criteria:

1. aged <18 years
2. pregnant
3. receiving any medications
4. any co morbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:Forced Expiratory Volume in 1 second (FEV1), (liters)
Forced Vital Capacity | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:Forced Vital Capacity (FVC), (liters)
Tiffenau index | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Tiffenau index (FEV1/FVC, FEV1%)
Peak Expiratory Flow | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Peak Expiratory Flow (PEF), (liters/second )
Maximal Expiratory Flow (MEF) | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Maximal Expiratory Flow (MEF) at 25%, 50%, and 75% of vital capacity,(liters/second )
Functional Residual Capacity (FRC) | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:Functional Residual Capacity (FRC), (liters)
Total Lung Capacity (TLC) | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Total Lung Capacity (TLC), (liters)
Residual Volume (RV) | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Residual Volume (RV), (liters)
Diffusion Capacity (DLCO) | 5 minutes after smoking IQOS
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Diffusion Capacity (DLCO) ((mmol/min/kPa)
Respiratory impedance | 5 minutes after smoking IQOS
  Total respiratory resistances measurement with an impulse oscillometry system (IOS)( (Viasys Jaeger MasterScreen IOS system) prior to smoking heated tobacco IQOS and 5 minutes after smoking IQOS were performed. The changes in:
  Respiratory impedance at 5 Hz (Z5Hz) (kPa/L/sec) were assessed
Total respiratory resistances | 5 minutes after smoking IQOS
  Total respiratory resistances measurement with an impulse oscillometry system (IOS)( (Viasys Jaeger MasterScreen IOS system) prior to smoking heated tobacco IQOS and 5 minutes after smoking IQOS were performed. The changes in:
  respiratory resistance at 5 (R5Hz),10 Hz (R10Hz),20 Hz (R20Hz) (kPa/L/sec) were assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Failure Unit, G Papanikolaou Hospital, Aristotle Unioversity of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No